CLINICAL TRIAL: NCT03619369
Title: Timing of Circumcision and Breastfeeding Frequency: A Randomized Clinical Trial
Brief Title: Circumcision and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Thornton Mu, Neonatologist, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C.2016.112d
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Breastfeeding, Exclusive; Circumcision
MeSH Terms: conditions — Breast Feeding | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Circumcision (Active Comparator)
  Interventions: Procedure: Circumcision
- Routine Circumcision (Placebo Comparator)
  Interventions: Procedure: Circumcision
- Delayed Circumcision (Active Comparator)
  Interventions: Procedure: Circumcision

INTERVENTIONS:
Procedure: Circumcision — Early vs. Routine vs. Delayed Circumcision and their impact on exclusive breastfeeding rates

SUMMARY:
1) To determine when the majority of male infants are being circumcised at 3 hospitals across the US (Brooke Army Medical Center, Naval Medical Center San Diego, and Dartmouth Hitchcock Medical Center. 2) To assess the breastfeeding patterns of circumcised male infants at the above-mentioned academic medical centers. Specifically, to determine if these babies are breastfeeding at the time of hospital discharge, at their newborn visit, their 2-week visit, and all subsequent well visits up until 6 months of age.

3) To determine if there is a significant relationship between the timing of newborn circumcision and breastfeeding initiation, establishment, and maintenance in the first 6 months of life. We hypothesize that the timing of circumcision will not be significantly associated with frequency of breastfeeding among mother-infant dyads during the initial months of life.

ELIGIBILITY:
Inclusion Criteria:

* All male infants born at the 3 participating sites

Exclusion Criteria:

* Gestational age <38 weeks, twin/multiple deliveries, NICU admission, mothers who are strictly formula feeding their newborns from the time of delivery, and mothers under 18 years of age.

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Rates | From birth thru 6 months of age
  Exclusive Breastfeeding Rates

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mondzelewski L, Mu T, Michalski A, Ward J, Cheng L, Chen M, Riffenburgh R, Holmes A. Timing of Circumcision and Breastfeeding Frequency: A Multicenter, Randomized Clinical Trial. Hosp Pediatr. 2022 Jun 1;12(6):555-560. doi: 10.1542/hpeds.2021-006400. PMID 35574656